CLINICAL TRIAL: NCT06825767
Title: Comparison of the Effectiveness of High-Intensity and Low-Intensity Laser Therapies in Primary Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nida Koçer Nazlıgül, Medical Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1-20-1087
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Primary Knee Osteoarthritis
Keywords: Osteoarthritis, Low level light therapy, high level light therapy,Muscle Skeletal; Ultrasonography
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- conventional treatment (Active Comparator): Conventional treatment including hotpack therapy, Transcutaneous Electrical Nerve Stimulation (TENS), joint range of motion exercises, straight leg lifting exercises, quadriceps strengthening exercises, pillow squeezing exercises, balance exercises on one leg for 4 weeks, 3 days a week for 4 weeks in 24 patients.
  Interventions: Device: Conventional Treatment
- conventional treatment and HILT(high-intensity laser therapy) (Active Comparator): Conventional treatment and HILT including hotpack therapy, Transcutaneous Electrical Nerve Stimulation (TENS), joint range of motion exercises, straight leg lifting exercises, quadriceps strengthening exercises, pillow squeezing exercises, balance exercises on one leg and HILT for 4 weeks, 3 days a week for 4 weeks in 24 patients .
  Interventions: Device: conventional treatment and high-intensity laser therapy(HILT)
- conventional treatment and LLLT(low-intensity laser therapy) (Active Comparator): Conventional treatment and LLLT including hotpack therapy, Transcutaneous Electrical Nerve Stimulation (TENS), joint range of motion exercises, straight leg lifting exercises, quadriceps strengthening exercises, pillow squeezing exercises, balance exercises on one leg and LLLT for 4 weeks, 3 days a week for 4 weeks in 24 patients.
  Interventions: Device: conventional treatment and low-intensity laser therapy (LLLT)

INTERVENTIONS:
Device: Conventional Treatment — Conventional treatment including hotpack therapy, Transcutaneous Electrical Nerve Stimulation (TENS), joint range of motion exercises, straight leg lifting exercises, quadriceps strengthening exercises, pillow squeezing exercises, balance exercises on one leg for 4 weeks, 3 days a week for 4 weeks in 24 patients
  Arms: conventional treatment
Device: conventional treatment and high-intensity laser therapy(HILT) — Conventional treatment and HILT including hotpack therapy, Transcutaneous Electrical Nerve Stimulation (TENS), joint range of motion exercises, straight leg lifting exercises, quadriceps strengthening exercises, pillow squeezing exercises, balance exercises on one leg and HILT for 4 weeks, 3 days a week for 4 weeks in 24 patients .
  Arms: conventional treatment and HILT(high-intensity laser therapy)
Device: conventional treatment and low-intensity laser therapy (LLLT) — Conventional treatment and LLLT including hotpack therapy, Transcutaneous Electrical Nerve Stimulation (TENS), joint range of motion exercises, straight leg lifting exercises, quadriceps strengthening exercises, pillow squeezing exercises, balance exercises on one leg and LLLT for 4 weeks, 3 days a week for 4 weeks in 24 patients.
  Arms: conventional treatment and LLLT(low-intensity laser therapy)

SUMMARY:
Our primary goal is to investigate the advantages of low-intensity laser therapy (LLLT) and high-intensity laser therapy (HILT) over conventional therapy in patients with knee osteoarthritis (OA), our secondary goal is to investigate the advantages of HILT and LLLT; to compare its analgesic effects, its effects on functional status and quality of life, and its effects on femoral cartilage thickness.

DETAILED DESCRIPTION:
In the study, those who applied to Ankara City Hospital Physical Therapy and Rehabilitation Hospital outpatient clinic between 01.10.2020-01.10.2021, were between the ages of 55-75, were diagnosed with primary knee OA according to the American Rheumatology Association, stage 2-3 knee according to Kellgren and Lawrence radiological classification. with OA; 72 volunteer patients with knee pain with a visual pain score of 4 and above for at least 3 months were included. The study was designed as a prospective, randomized, controlled, single-center. Patients were randomly divided into 3 treatment groups. Conventional treatment including hotpack therapy, Transcutaneous Electrical Nerve Stimulation (TENS), joint range of motion exercises, straight leg lifting exercises, quadriceps strengthening exercises, pillow squeezing exercises, balance exercises on one leg for 4 weeks, 3 days a week for 4 weeks in 24 patients in the first group, conventional treatment and HILT were applied to 24 patients in the second group, and conventional treatment and LLLT were applied to 24 patients in the third group. All groups were evaluated clinically and ultrasonographically at the beginning of the treatment, at the end of the treatment and at the 3rd month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 55-75 years
* Primary knee OA diagnosis according to ACR (American College of Rheumatology) and Knee OA classified as stage 2-3 according to the KL (Kellgren-Lawrence) radiological classification
* Visual pain score of 4 or higher for knee pain lasting for at least 3 months

Exclusion Criteria:

* Patients with secondary knee OA
* Patients who have undergone surgical operations related to the knee joint
* Patients with pathology in the hip and/or ankle on the same side
* Patients who have received intra-articular corticosteroid, hyaluronic acid, or PRP injections in the knee joint in the last 6 months
* Patients who have received physical therapy for the knee region in the last 6 months
* Patients with serious systemic diseases such as malignancy, congestive heart failure, or chronic obstructive pulmonary disease
* Patients with insufficient cognitive function

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
range of motion | Baseline, after 1 month and 3 month changes
  In the clinical evaluation, the range of motion of the patients in the affected extremity was determined by goniometry
visual pain score (VAS) | Baseline, after 1 month and 3 month changes
  In the clinical evaluation, the pain score with movement and resting was determined by visual pain score (VAS).The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, after 1 month and 3 month changes
  Western Ontario and McMaster Universities (WOMAC) index is the most common used clinical tools for evaluating patients with knee OA.It is consisted of 33 items which evaluates the health and function of the patient from various aspects including: clinical symptoms (5 questions), severity of joint stiffness (2 questions), degree of pain (9 questions), and activity of daily living (17 questions).
  Each question has five subscales where best situation scores as never or none and the worst one names as extreme or always. Here, higher scores are representative of better situation and less pain.
Lequesne Index | Baseline, after 1 month and 3 month changes
  The Lequesne index has an interview format questionnaire, including 10 questions divided into three sections regarding pain, maximum distance walked and activities of daily living . The score ranges from 0 (no pain, no disability) to 24 (maximum pain and disability
Short form SF-36 scale | Baseline, after 1 month and 3 month changes
  The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.
Femoral cartilage thickness | Baseline, after 1 month and 3 month changes
  The femoral cartilage thickness measurements of the patients participating in the study were performed using a Logiq 9 (GE Medical Systems®) ultrasound device with a linear probe (7-12 MHz, "ZONARE"). The ultrasonographic measurement was performed in the supine position of the patient, with the knee in maximum flexion, at three different locations: the medial femoral intercondylar region, the median intercondylar region, and the lateral femoral intercondylar region. The probe was placed transversely on the thigh, perpendicular to the bone surface, immediately above the superior corner of the patella. The cartilage thickness was calculated by measuring the hypoechoic distance between the two hyperechoic lines: one showing the soft tissue-cartilage surface and the other showing the cartilage-bone surface. Three measurements were taken for each knee, and the average was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital Phisical Therapy and Rehabilitation Hospital, Ankara, Bilkent-Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No